CLINICAL TRIAL: NCT04158310
Title: Evaluation of Clinical Value and Safety of Xiyanping Injection in the Treatment of Community-acquired Pneumonia in Children Based on Real-world Clinical Data
Brief Title: Evaluation the Clinical Value of Xiyanping Injection in the Treatment of Community-acquired Pneumonia in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QF-XYP1908-2
Record Dates: First submitted 2019-10-30; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard treatment only: Standard treatment only such as antiasthmatic, expectorant and antipyretic
- Standard treatment+Xiyanping injection: Standard Treatment such as antiasthmatic, expectorant and antipyretic plus Xiyanping injection intravenous administration of 0.2-0.4mL/kg/day ,QD.

SUMMARY:
In order to verify the clinical value and safety of Xiyanping injection in children with CAP, we intend to carry out this multi-center, large-sample, non-intervention clinical research through more rigorous and scientific design. Considering the current status of clinical research in children in China,research use real-world research methods.

DETAILED DESCRIPTION:
This is an real world study of efficacy and safety of intravenous injection of Xiyanping injection in pediatric subjects with CAP.The purpose to determine the clinical value and influencing factors of Xiyanping injection in the treatment of community-acquired pneumonia in children based on real-world clinical data. The starting point for the study was the time at which the patient started treatment with Xiyanping injection or using a conventional treatment regimen; the end of follow-up was the date of the last visit to the patient, and if the patient had a disease progression or transfer, the date of the occurrence was the end. At the same time, baseline demographic characteristics (gender, date of birth, type of medical insurance, etc.), therapeutic drugs during the follow-up period, dose and time of use, laboratory indicators (such as white blood cells, C-reactive protein, etc., and examination time) were collected.

ELIGIBILITY:
Inclusion criteria:

* 2 years old < age ≤ 14 years old children, male or female, diagnosed as community-acquired pneumonia diagnosed and need hospitalization

Exclusion criteria:

* Acute infectious diseases such as measles, whooping cough, and influenza
* Other concomitant diseases or conditions that the investigators believe may interfere with the study, such as severe primary disease with severe heart, liver, kidney, digestive, and hematopoietic systems
* Children with severe malnutrition and previous history of immunodeficiency may seriously affect the self-limiting course of the disease
* Children with epilepsy and other central nervous system dysfunction
* Congenital diseases, mental patients
* Those who have used systemic hormones within 2 weeks before enrollment;
* Those who have used Qingrejiedu Chinese medicine within 2 weeks before enrollment
* The subject is poorly compliant (not according to the doctor's prescription or medical advice) or fails to timely feedback information

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2 years old < age ≤ 14 years old children, male or female, diagnosed as community-acquired pneumonia diagnosed and need hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 9207 (Estimated)
Dates: Start 2019-11-11 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to Alleviation of Cough and Lung X-ray | 7 days
  significant efficiency: cough and lung X-ray show obvious improvement of symptoms within 3 days; effective: cough and lung X-ray symptoms improve within 3 to 7 days; invalid: no change or aggravation of lung symptoms after 7 days' treatment. Total effective rate = significant efficiency rate + effective rate
Time to Alleviation of Body Temperature | 7 days
  significant efficiency: body temperature return to normal within 3 days; effective: body temperature return to normal within 3 to 7 days; invalid: body temperature can't return to normal after 7 days' treatment. Total effective rate = significant efficiency rate + effective rate